CLINICAL TRIAL: NCT03136510
Title: Prospective Study With Biological Assessment: Evolution of Coagulation Activity in Non Valvular Atrial Fibrillation Patients Under Apixaban
Brief Title: Evolution of Coagulation Activity in Non Valvular Atrial Fibrillation Patients Under Apixaban
Acronym: ECAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Dr Jean-Guillaume DILLINGER, Jean Guillaume DILLINGER, MD,PhD, principal investigator, Hopital Lariboisière
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CV185-439
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2019-03

CONDITIONS: Coagulation Disorder; Non Valvular Atrial Fibrillation
MeSH Terms: conditions — Hemostatic Disorders | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: 60 patients with two subgroups
  * 30 patients with new diagnosis of atrial fibrillation (vitamin K antagonist treatment shorter than 1 week) : initiated with Apixaban 5 mg
  * 30 patients previously chronically treated by VKA for more than 3 months and switched to Apixaban 5 mg
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newly diagnosed NVAF: apixaban 5 mg (Other): blood collection for biological analyses of 30 patients new diagnosis of NVAF (VKA treatment ≤1 week) initiated with apixaban 5 mg
  Interventions: Drug: Apixaban 5 mg
- Previously diagnosed NVAF: apixaban 5 mg (Other): blood collection for biological analyses of 30 patients previously treated by VKA for more than 3 months switched to apixaban 5 mg
  Interventions: Drug: Apixaban 5 mg

INTERVENTIONS:
Drug: Apixaban 5 mg — Bood collection for biological analyses at:
  * inclusion visit
  * follow-up visit at 1 month
  * end of research at 3 month
  Other Names: Eliquis

SUMMARY:
Apixaban is a potent, oral, selective reversible direct inhibitor of factor Xa with a favorable efficacy and safety profile in the prevention of non valvular (NV) atrial fibrillation (AF). It has been shown, including by our group, that D-dimers levels (molecular marker of coagulation activity) are predictive of the events (including mortality) in patient with AF independently of the antithrombotic treatment. The aim of the study is to evaluate the changes in plasma levels of biomarkers of coagulation activation: D-dimers, prothrombin fragments F1+2, von Willebrand factor (vWF) and thrombin-antithrombin complexes (TAT) in response to apixaban treatment in patients with NVAF.

DETAILED DESCRIPTION:
This study is a prospective, monocentric study, with biological analyses. The investigational product will be administered according to French health agency. The duration of the study for each patient will be 3 months with 3 visits and from 3 to a maximum of 18 months for the clinical follow-up.

Hypothesis: Apixaban significantly decreases D-dimers and other markers of coagulation activation in patients with NVAF ( paroxysmic and chronic atrial fibrillation).

Primary endpoint:

Measurement of D-dimers at baseline (before apixaban treatment) and under chronic apixaban treatment at 3 months in the overall population.

Secondary endpoints:

Difference of the D-dimers levels between enrollment (V1) and the final visit (V3) at three months in both subgroups separately. In the subgroup B,comparison of D-dimers in patients previously treated by VKA (V1) and under apixaban (V3).

Similarly than for D-dimers levels, each following parameters will be analyzed for the overall population and for both subgroups separately :

* Difference of prothrombin fragments F1+F2 levels between V1 and V3.
* Difference of thrombin and antithrombin complexes levels between V1 and V3
* Difference of vWF levels between V1 and V3.

Correlation will be evaluated between:

* AntiXa apixaban activity (at trough) and D-dimers difference
* D-dimers difference and clinical follow-up (ischemic events and-bleeding events) V2 and V3 levels of each parameter will be compared to assess the delay of appearance of the apixaban effect if any. Inflammation parameters ( C reactive protein and fibrinogen) will be used as explicative for the other parameters.

Effect on APTT( activated partial thromboplastin time) and PT(prothrombin time) will be compared to specific apixaban anti Xa activity

Subgroup analysis:

* Subgroups A and B (newly diagnosed and VKA naïve NVAF and chronic NVAF)
* age >80 years,
* creatinine clearance < 50 ml/min,
* gender Multivariate analysis for the primary endpoint

Statistical analysis Continuous variables will be analyzed for a normal distribution with the D'Agostino-Pearson test. They will be presented as mean and standard deviation (SD) and compared with Student's unpaired t-test if normally distributed, or presented as median and interquartile range and compared with Mann-Whitney rank-sum test, if not. Categorical variables will be presented as counts and percentages and will be compared by means of the χ2-test or Fisher's exact test.

Correlations between quantitative variables will be assessed with Pearson correlation coefficients. Predictive factors will be determined using a stepwise multivariable logistic regression analysis. In this study, we will expect an initial D-dimers level around 1500ng/ml with a standard deviation of ±700ng/ml in patients with newly diagnosed NVAF. At 3 month, we expect a level of D-dimers of 1000±600ng/ml (reduction of 500ng/ml compared to the enrolment visit). A sample size of 60 patients has been estimated in this pilot study. The study will include 60 patients with NVAF with 50% of patients with newly diagnosed NVAF (Subgroup A, n=30) and the other 50% with NVAF previously treated by VKA (Subgroup B, n=30).

All information required by the protocol must be provided in the case report form. The data will be transferred in the case report forms as and when they are obtained, whether clinical or biological. The investigators will make the data available strictly necessary for qua lity control and audit relating to the biomedical research in accordance with the legislative and regulatory provisions in force (Articles L.1121-3 and R.5121-13 of the French Public Health Code).

Those responsible for biomedical research quality control (Article L.1121-3 of the French Public Health Code) will take all necessary precautions to ensure the confidentiality of information about the experimental medications, the research, the research subjects and in particular the identity of the subjects and the results obtained. These individuals, as well as the investigators themselves, are subject to professional secrecy (in accordance with the conditions set out in Articles 226-13 and 226-14 of the Penal Code).

All Serious Adverse Events (SAEs) that occur following the subject's written consent to participate in the study through 30 days of discontinuation of dosing must be reported to Bristol-Myers Squibb Worldwide Safety and to the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NVAF (documented by 12 leads ECG or Holter recording) and having one or more factor (s) of risk such as: history of stroke or transient ischemic attack ; age≥75 years; hypertension; diabetes; symptomatic heart failure (NYHA class≥ II) for prevention of cerebral vascular accident and systemic embolism.
* Patients with CHA2DS2-VASc score ≥2
* Patients provided signed written informed consent
* Patients with age≥18 years
* Patients previously treated with VKA or patients newly diagnosed with AF.

Exclusion Criteria:

* AF or flutter due to reversible causes according to investigator
* Clinically significant mitral stenosis
* Any other condition than atrial fibrillation that require chronic anticoagulation (prosthetic heart valve or valve repair, venous thromboembolism)
* A need for aspirin at a dose of ≥160 mg a day or for both aspirin and adenosine diphosphate (ADP) inhibitor (clopidogrel, prasugrel or ticagrelor)
* Allergy or adverse reaction to apixaban or any of the excipients
* Patients previously treated by an oral direct anticoagulant in the last 30 days
* Patient with clinically on going active bleeding or platelet count<100,000/mm3 or haemoglobin<9 g/dL
* Patients with serious bleeding in the last 6 months or with high risk of bleeding (active peptic ulcer disease or gastroduodenal ulceration, known or suspected esophageal varicoses, recent ischemic stroke, recent brain or spinal injury or intracranial hemorrhage, recent surgery, arterial or venous malformations, vascular aneurysms…)
* Patients with another cause of increase of D-dimers (active malignant neoplasm, recent trauma or surgery (less than 1 month), extensive venous malformation…)
* Uncontrolled and persistent hypertension (systolic >180 mmHg or diastolic >100 mmHg)
* Active infective endocarditis
* aspartate transaminase (ASAT) or alanine aminotransferase (ALAT) > 2 times upper limit or hepatic disease with coagulopathy
* Severe renal insufficiency (creatinine clearance <30ml/min)
* Women in age of pregnancy without menopause or efficient contraception and pregnant women or breast feeding women. Men without effective contraception.
* Any reason that makes the study participation impractical (alcohol abuse, psychosocial reason, inclusion in another study in the past month, life expectancy≤1 year…)
* Any contraindications to study treatment (apixaban): hypersensitivity to apixaban or any of the excipients (see composition), ongoing active bleeding, hepatic disease with coagulopathy, any condition with high risk of bleeding, concomitant anticoagulant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
change from baseline D-dimers level at 3 months. | 3 months
  D-dimers levels will be determined using an enzyme immunoassay (ELISA method) on citrated plasma.

SECONDARY OUTCOMES:
Prothrombin fragment F1-F2 measurement | at enrollment, at one month, and at three months
  Prothrombin fragment F1-F2 will be determined using an enzyme immunoassay (ELISA method) on citrated plasma.
von Willebrand factor measurement | at enrollment, at one month, and at three months
  vWF will be determined using an enzyme immunoassay (ELISA method) on citrated plasma.
Thrombin-antithrombin complex measurement | at enrollment, at one month, and at three months
  TAT complex will be determined using an enzyme immunoassay (ELISA method) on citrated plasma.
High sensitivity CRP measurement | at enrollment, at one month, and at three months
  Hs CRP will be measured following usual method of the biochemistry laboratory on EDTA (ethylenediaminetetraacetic acid ) plasma.
Prothrombin time measurement, Activated partial thromboplastin time, and fibrinogen | at enrollment, at one month, and at three months
  Prothrombin time, a PTT and fibrinogen will be measured following usual method of the hematology laboratory on citrated plasma.
AntiXa apixaban activity measurement | at enrollment, at one month, and at three months
  Anti-Xa apixaban levels will be determined using the specific technic with adapted apixaban calibrators on citrated plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic DROUET, MD, PhD, Study Director — Lariboisiere Hospital
Locations (1):
- Department of Cardiology Lariboisiere Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No